CLINICAL TRIAL: NCT00092703
Title: A Randomized, Double-Blind, Multicenter Study to Evaluate the Tolerability and Effectiveness of Etoricoxib 90 mg q.d. vs. Diclofenac Sodium 50 mg t.i.d. in Patients With Osteoarthritis
Brief Title: Investigational Drug Versus an Approved Drug in Patients With Osteoarthritis (0663-061)(COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0663-061; 2004_052
Record Dates: First submitted 2004-09-23; First posted 2004-09-28 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2022-02

CONDITIONS: Osteoarthritis
Keywords: Arcoxia
MeSH Terms: conditions — Osteoarthritis | interventions — Etoricoxib

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: MK0663, etoricoxib
Drug: Comparator: Diclofenac sodium

SUMMARY:
The purpose of this study is to compare the gastrointestinal tolerability of an investigational drug to an approved drug in the treatment of osteoarthritis during one year treatment period.

DETAILED DESCRIPTION:
The duration of treatment is 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Osteoarthritis of the knee, hip, hand or spine which requires the use of medications for pain relief

Exclusion Criteria:

* Known allergies to the study drugs

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6000
Dates: Start 2002-06-27 (Actual); Primary Completion 2003-11-01 (Actual); Study Completion 2003-11-01 (Actual)

PRIMARY OUTCOMES:
Discontinuations due to clinical and laboratory gastrointestinal adverse experiences during a 1 year treatment period.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Baraf HS, Fuentealba C, Greenwald M, Brzezicki J, O'Brien K, Soffer B, Polis A, Bird S, Kaur A, Curtis SP; EDGE Study Group. Gastrointestinal side effects of etoricoxib in patients with osteoarthritis: results of the Etoricoxib versus Diclofenac Sodium Gastrointestinal Tolerability and Effectiveness (EDGE) trial. J Rheumatol. 2007 Feb;34(2):408-20. PMID 17304660
- [Background] Cannon CP, Curtis SP, FitzGerald GA, Krum H, Kaur A, Bolognese JA, Reicin AS, Bombardier C, Weinblatt ME, van der Heijde D, Erdmann E, Laine L; MEDAL Steering Committee. Cardiovascular outcomes with etoricoxib and diclofenac in patients with osteoarthritis and rheumatoid arthritis in the Multinational Etoricoxib and Diclofenac Arthritis Long-term (MEDAL) programme: a randomised comparison. Lancet. 2006 Nov 18;368(9549):1771-81. doi: 10.1016/S0140-6736(06)69666-9. PMID 17113426
- [Background] Laine L, Curtis SP, Cryer B, Kaur A, Cannon CP; MEDAL Steering Committee. Assessment of upper gastrointestinal safety of etoricoxib and diclofenac in patients with osteoarthritis and rheumatoid arthritis in the Multinational Etoricoxib and Diclofenac Arthritis Long-term (MEDAL) programme: a randomised comparison. Lancet. 2007 Feb 10;369(9560):465-73. doi: 10.1016/S0140-6736(07)60234-7. PMID 17292766
- [Background] Krum H, Curtis SP, Kaur A, Wang H, Smugar SS, Weir MR, Laine L, Brater DC, Cannon CP. Baseline factors associated with congestive heart failure in patients receiving etoricoxib or diclofenac: multivariate analysis of the MEDAL program. Eur J Heart Fail. 2009 Jun;11(6):542-50. doi: 10.1093/eurjhf/hfp054. Epub 2009 Apr 19. PMID 19380329
- [Background] Laine L, Curtis SP, Langman M, Jensen DM, Cryer B, Kaur A, Cannon CP. Lower gastrointestinal events in a double-blind trial of the cyclo-oxygenase-2 selective inhibitor etoricoxib and the traditional nonsteroidal anti-inflammatory drug diclofenac. Gastroenterology. 2008 Nov;135(5):1517-25. doi: 10.1053/j.gastro.2008.07.067. Epub 2008 Aug 3. PMID 18823986
- [Background] Laine L, Goldkind L, Curtis SP, Connors LG, Yanqiong Z, Cannon CP. How common is diclofenac-associated liver injury? Analysis of 17,289 arthritis patients in a long-term prospective clinical trial. Am J Gastroenterol. 2009 Feb;104(2):356-62. doi: 10.1038/ajg.2008.149. Epub 2009 Jan 27. PMID 19174782